CLINICAL TRIAL: NCT04118998
Title: Progressive Abduction Loading Therapy: A Phase IIb Stroke Rehabilitation Trial With Longitudinal Tracking
Brief Title: Progressive Abduction Loading Therapy
Acronym: PRALINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Shirley Ryan AbilityLab (Other); Marianjoy Rehabilitation Hospital & Clinics (Other)
Responsible Party: Principal Investigator, Michael Ellis, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00209671; R01HD096071 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stroke, Acute
Keywords: Rehabilitation; Arm; Flexion Synergy; Longitudinal; Targetted; Quantitative
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two arms or study interventions are indistinguishable by patients and untrained observers. The Care Providers (Study Intervention Therapists) can not be masked due to their knowledge in the delivery of the physical intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abduction Loading (Experimental): The intervention for the experimental group entails practicing reaching with abduction loading.
  Interventions: Behavioral: Abduction Loading
- Supported Reaching (Active Comparator): The intervention for the active comparator entails practicing reaching while supported.
  Interventions: Behavioral: Supported Reaching

INTERVENTIONS:
Behavioral: Abduction Loading — The intervention for the experimental group entails practicing reaching with abduction loading.
  Other Names: Progressive Abduction Loading Therapy
  Arms: Abduction Loading
Behavioral: Supported Reaching — The intervention for the active comparator entails practicing reaching while supported.
  Arms: Supported Reaching

SUMMARY:
This study attempts to minimize the development of a common movement impairment following stroke known as "flexion synergy" that makes it extremely difficult to reach outward with the arm. Participants with acute/subacute stroke will receive one of two study interventions in addition to prescribed therapies in both inpatient rehabilitation and day-rehab. Participants will be followed for 1 year.

DETAILED DESCRIPTION:
Eighty-six individuals with acute (admission to in-patient rehabilitation) severe hemiparetic stroke (Chedoke McMaster Stroke Assessment arm score of Stage 2 or 3 out of 7) will participate in this study. All participants will be recruited upon admission to the Shirley Ryan AbilityLab (formally Rehabilitation Institute of Chicago) for stroke rehabilitation under the administration of the study physician. Participants will receive experimental or comparison group therapy as adjuvant to regular in-patient and day-rehabilitation therapy. Participants will be evaluated weekly while in therapy and then bimonthly (every other month) after discharge until 1-year following baseline evaluation.

From the admission evaluations by the study physician and other rehabilitation services, patients with adequate language, visuospatial, cognitive and motor function will be consented for participation and then screened by a study evaluation physical therapist and board-certified neurological clinical specialist for the specific motor inclusion criteria. After consent, a REDCap screening form will be initiated by the study physician's project coordinator with relevant data from the participant medical record. The study evaluation therapist will then conduct the screening that will include verification and completion of the inclusion/exclusion criteria and the transcranial magnetic stimulation (TMS) safety checklist that will identify any contraindication to TMS-based assessment of motor evoked potentials (MEPs). The Chedoke McMaster Stroke Assessment (primary motor inclusion criteria) is very time efficient reducing interference with in-patient therapy activities and rapidly identifying individuals with severe impairment facilitating participant recruitment. The study evaluation therapist will not need to complete the entire assessment instead only confirming patients at level 2 and 3 out of 7 for inclusion. The REDCap screening form and TMS checklist will be reviewed by the study physician. The study physician will grant medical clearance for TMS-based MEP assessment and participation in the study.

Regarding motor criteria; participants not meeting the minimum of Stage 2 out of 7 on the Chedoke McMaster Stroke Assessment will be monitored for emergence of adequate movement. Shirley Ryan AbilityLab therapists routinely report Chedoke scores in daily documentation. The study physician and project coordinator will notify the study evaluation therapist once minimal movement emerges in these patients and the screening process can be initiated. Participants who subsequently pass screening and medical clearance for TMS-based MEP assessment will undergo conventional MEP assessment. Participants will later be randomly allocated to either the experimental or comparison treatment groups within REDCap by the study intervention therapist upon the first intervention session. The REDCap randomization algorithm is managed by the study biostatistics team and employs a concealed allocation table. The allocation table is constructed to balance the allocation of participants (2 groups of n=43) by sex, presence or absence of MEPs, and level of severity as measured by the Fugl-Meyer Arm Motor Assessment in order to ensure equivalent baseline characteristics of each group. The Fugl-Meyer score will be divided in bins of 6 points. Participants, evaluation therapists, biostatisticians, and the study PD/PI will be blinded to group assignment. Intervention therapists and the study physician will not be blinded to group assignment. Participants will not be able to tell the difference between interventions since both will involve reaching practice. Participants that are not medically cleared for TMS-based MEP assessment will be randomly allocated to group without MEP status. It is anticipated that only 1-2% of participants will not be cleared for MEP assessment.

Baseline and subsequent evaluations will include a kinematic/kinetic measurement of reaching function (primary endpoint, reaching distance under standardized abduction loading, normal gravity) and a kinematic/kinetic measurement of shoulder/elbow impairment (secondary endpoint, loss of independent joint control). The primary and secondary endpoints will be conducted at Shirley Ryan AbilityLab during both in-patient and day-rehabilitation by the study evaluation therapist under following initial training and certification by the study PD/PI. Standardized clinical evaluations of arm impairment, activity limitation, and participation restriction will also be performed during this phase at Shirley Ryan AbilityLab by the study evaluation therapist who will be blinded to intervention group. Evaluations will take place at baseline, weekly until discharge from rehabilitation, and then bimonthly until 12 months post-baseline measurement. Following discharge from rehabilitation, patients will receive follow-up evaluations bimonthly at Northwestern University Department of Physical Therapy and Human Movement Sciences. These evaluations will be conducted by a second study evaluation therapist and board-certified neurological clinical specialist following initial training and certification by the study PD/PI. The second study evaluation therapist will also serve as the backup for the first study evaluation therapist in case of illness/absence.

During in-patient rehabilitation and day-rehabilitation, experimental and comparison intervention sessions will parallel regular therapy and be conducted at Shirley Ryan AbilityLab and Streeterville Day Rehabilitation Center respectively by two Shirley Ryan AbilityLab study intervention therapists. Study intervention therapists will be initially trained and certified by the study PD/PI. Study intervention sessions will be 5 days per week during in-patient therapy and 3 days per week during day-rehabilitation. The intervention period for both groups will be ~45 minutes (truncated at 1 hour) in addition to the regular therapy schedule until discharge. Both interventions will involve performing standardized reaching exercises to outward targets displayed on a monitor. The experimental group receiving progressive abduction loading therapy will practice reaching exercises with abduction loading and the comparison group will practice reaching supported on a horizontal haptic table. All participants will have the same maximum number of sets and repetitions of exercise during sessions and the sessions will be truncated at 60 minutes of total contact time. Half of the enrolled participants are expected to transition to day-rehabilitation following in-patient rehabilitation. In day-rehabilitation, participants will continue to receive the same study intervention but only 3 days per week matching the day-rehabilitation schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Hemiparesis confined to one side, (CMSA Stage 2 or 3 out of 7)
2. Stroke impacting parenchyma of the middle cerebral artery distribution
3. Within 90 days post-stroke
4. 18 to 85 years old
5. No or Mild-to-moderate Aphasia (NIHSS #9 Best Language. = 0 or 1- Describe picture; No or Mild-to-moderate Aphasia)
6. No or Mild extinction and inattention (NIHSS 11 Extinction and Inattention. = 0 or 1- No abnormality or Inattention to one modality.)
7. Ability to perform a 3-step motor command with the unaffected arm
8. Capacity to provide informed consent

Exclusion Criteria:

1. Premorbid and persistent disability or motor impairment of the upper extremities
2. Brainstem and/or cerebellar lesion
3. Comorbidity medically contraindicating motor assessments
4. Any other chronic neurological condition
5. Pain or hypersensitivity limiting motor assessments
6. Limb edema limiting study motor assessments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Reaching Function | Change in Reaching function will be modeled from baseline, weekly (until discharge from rehabilitation, on average 4 to 10 weeks), and monthly evaluations (every-other month until 12 months post-stroke).
  Quantitative evaluation of reaching by calculating distance from reaching kinematics data during ballistic outward reaches against gravity.

SECONDARY OUTCOMES:
Change in Loss of Independent Joint Control | Change in Loss of Independent Joint Control will be modeled from baseline, weekly (until discharge from rehabilitation, on average 4 to 10 weeks), and monthly evaluations (every-other month until 12 months post-stroke).
  Quantitative evaluation of the expression of flexion synergy impairment. Measured as the maximum abduction load achieved during a reach to two standardized targets (near and far).
Change in Fugl-Meyer Motor Assessment | Change in Fugl-Meyer Motor Assessment will be modeled from baseline, weekly (until discharge from rehabilitation, on average 4 to 10 weeks), and monthly evaluations (every-other month until 12 months post-stroke).
  Qualitative and clinical assessment of general motor impairment of arm following stroke. The scale evaluates movement impairment of the arm through observation. The scale ranges from 0-66 points with 66 indicating the best score.
Change in Action Research Arm Test | Change in Action Research Arm Test will be modeled from baseline, weekly (until discharge from rehabilitation, on average 4 to 10 weeks), and monthly evaluations (every-other month until 12 months post-stroke).
  Qualitative and clinical assessment of activity limitation (function) of the arm following stroke. The scale focusses on reaching, grasping, and releasing objects of various sizes. The scale ranges from 0-57 with 57 indicating the best score.
Change in Stroke Impact Scale | Change in Stroke Impact Scale will be modeled from baseline, weekly (until discharge from rehabilitation, on average 4 to 10 weeks), and monthly evaluations (every-other month until 12 months post-stroke).
  Structured interview to assess domains of the ICF (International Classification of Functioning, Disability and Health) in individuals following stroke. The domains include self-reported physical problems, memory and thinking, control of emotions, communication, daily activities, home and community mobility, the affected hand, participation and life roles, and global recovery. Each domain score is transformed to a scale of 0-100 with 100 being the best score.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Ellis, PT, DPT, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Northwestern Medicine Marianjoy Rehabilitation Hospital, Wheaton, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Final research data will be shared openly and timely in accordance with NIH Data Sharing Policy (https://grants.nih.gov/grants/policy/data_sharing/) and NICHD Data and Specimen Hub - Data Archive Policy Statement (https://dash.nichd.nih.gov/Resource/Policies). Data sharing will occur through the primary repositories of NICHD DASH (https://dash.nichd.nih.gov/), Northwestern University DigitalHub (https://digitalhub.northwestern.edu/), and Open Science Framework (https://osf.io/). Data will be exported from the internal RedCap study data base in spreadsheet format and will be deidentified and coded. Data will be available through speaking engagements and publications, presentations at scientific symposia and seminars. Data sharing in the above repositories will be phased in time with acceptance for publication of the primary outcome paper near the end of the fifth year and then with each subsequent publication. Publications will include DOIs for the data repositories.
Time Frame: Data sharing in the above repositories will be phased in time with acceptance for publication of the primary outcome paper near the end of the fifth year and then with each subsequent publication.
Access Criteria: Data sharing will occur through the primary repositories of NICHD DASH (https://dash.nichd.nih.gov/), Northwestern University DigitalHub (https://digitalhub.northwestern.edu/), and Open Science Framework (https://osf.io/). Data will be exported from the internal RedCap study data base in spreadsheet format and will be deidentified and coded. Data will be available through speaking engagements and publications, presentations at scientific symposia and seminars.
URL: http://dash.nichd.nih.gov/

REFERENCES:
- [Background] Yamada K. The glossophyaryngeal nerve response to taste and thermal stimuli in the rat, rabbit and cat. Kumamoto Med J. 1965 Jun 30;18(2):106-8. No abstract available. PMID 5825888
- [Background] Martig J, Riser WH, Germann F. Deforming ankylosis of the coffin joint in calves. Vet Rec. 1972 Sep 23;91(13):307-10. doi: 10.1136/vr.91.13.307. No abstract available. PMID 5086410
- [Background] Chou MY, Malison MD. Outbreak of acute hemorrhagic conjunctivitis due to coxsackie A24 variant--Taiwan. Am J Epidemiol. 1988 Apr;127(4):795-800. doi: 10.1093/oxfordjournals.aje.a114861. PMID 2833097
- [Derived] Roth HR, Carmona C, Clark G, Gyarmaty JE, Dewald JPA, Giblin E, Harvey RL, Jaskiewicz J, Kim KA, Lancki N, Luhrsen A, Mandana A, Manikonda D, Morris A, Sheth S, Stoykov ME, Young AC, Zielke D, Ellis MD. PRALINE: study protocol for a phase IIb inpatient stroke rehabilitation randomized controlled trial investigating longitudinal outcomes after progressive abduction loading therapy. Trials. 2025 Jul 20;26(1):250. doi: 10.1186/s13063-025-08969-6. PMID 40685355